CLINICAL TRIAL: NCT01429818
Title: Endothelial Disfunction Treatment With Glimepiride/Metformin Combination (Glimetal) in Type 2 Diabetes Patients. Positron Emission Tomography Assessment(PET)
Brief Title: Endothelial Disfunction Treatment With Glimepiride/Metformin Combination (Glimetal) in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PET-GLI01
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Endothelial Dysfunction; Diabetes Mellitus
Keywords: Endothelial dysfunction; Diabetes mellitus; glimepiride; metformin
MeSH Terms: conditions — Diabetes Mellitus | interventions — glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride/metformin (Experimental)
  Interventions: Drug: Glimepiride/metformin
- Metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Glimepiride/metformin — 4/1000 mg tablets once a day foe eight weeks
  Other Names: GLIMETAL
  Arms: Glimepiride/metformin
Drug: Metformin — 1000 mg tablets once daily for eight weeks
  Other Names: PREDIAL
  Arms: Metformin

SUMMARY:
The Purpose of this study was to evaluate the effect of the combination glimepiride/metformin over endothelial dysfunction (ED) in asymptomatic patients with type 2 diabetes mellitus (DM) using 13N-ammonia-positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* At least 18 years old
* Type 2 diabetes mellitus diagnosis
* Signed Informed Consent

Exclusion Criteria:

* History of smoking, hypertension, dyslipidemia, ischemic heart disease or autoimmune rheumatic diseases
* Pregnancy or lactation
* History of abuse and/or substance dependence within 6 months preceding the survey.
* History of glimepiride or metformin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
EDVI | 8 weeks
  endothelial-dependent vasodilation index
MFR | 8 weeks
  myocardial flow reserve
%ΔMBF | 8 weeks
  percentage of the change between rest and CPT

SECONDARY OUTCOMES:
Fasting glucose | 8 weeks
Glycated hemoglobin | 8 weeks
Adverse effects | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jorge González, MD, Study Director — Laboratorios Silanes S.A. de C.V.
Locations (1):
- Unidad PET Ciclotrón. Facultad de Medicina. Universidad Nacional Autónoma de México, Mexico City, Mexico City, Mexico